CLINICAL TRIAL: NCT02934841
Title: Conbercept in Choroidal Neovascularization Secondary to Uveitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Shulin Liu, Director, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BQE-10
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Choroidal Neovascularization; Uveitis
MeSH Terms: conditions — Choroidal Neovascularization; Uveitis | interventions — KH902 fusion protein; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conbercept (Experimental): The patients are followed on a monthly basis until 12 months. Three intravitreal injections of conbercept at a dosage of 0.5 mg are initiated at inclusion (monthly) with reinjection every month only in case of CNV activity (PRN regimen) until 12 months.
  Interventions: Drug: Conbercept
- sham (Sham Comparator): The patients are followed on a monthly basis until 12 months. Three intravitreal sham injections are initiated at inclusion (monthly) with reinjection every month only in case of CNV activity (PRN regimen) until 12 months.
  Interventions: Drug: sham

INTERVENTIONS:
Drug: Conbercept
  Arms: Conbercept
Drug: sham
  Arms: sham

SUMMARY:
The investigators hypothesize that it is safe and effective to treat patients with choroidal neovascularisation (abnormal blood vessels growing under the retina) secondary to uveitis with Conbercept.

This will be a randomized, placebo-controlled trial. 20 patients will receive three injections of Conbercept into the affected eye (and repeated injections if required), and 20 patients will receive three sham injections requiring no needle stick, but making the patient unaware of whether or not he received active treatment.

Outcome of the two treatment groups will be compared after one year.

DETAILED DESCRIPTION:
Primary Outcome Measures: Mean change from baseline in best corrected visual acuity [ Time Frame: 12 months ]

Secondary Outcome Measures: Mean change from baseline in retinal thickness [ Time Frame: 12 months ]

Mean number of Conbercept injections required over 12 months [ Time Frame: 12 months ]

Ocular and systemic adverse events [ Time Frame: 12 months ]

Enrollment: 40

Intervention Details: Drug: Conbercept

20 patients will receive an intravitreal injections of conbercept 0.5 mg at baseline (visit 1; month 0) then a subsequent intravitreal injection at month 1 (visit 2) and month 2 (Visit 3). Patients will be reviewed every month thereafter for 12 months at which time it will be determined whether the patient requires retreatment with conbercept 0.5 mg based on measurements of visual acuity, Optical coherence tomography (OCT) findings, FFA and clinical appearance.

ELIGIBILITY:
Inclusion Criteria:

* Patient with uveitis (without signs of active uveitis) related CNV, whatever the cause, including multifocal choroiditis, punctate inner choroidopathy, ocular toxoplasmosis, serpiginous choroiditis, Birdshot chorioretinopathy or VKH syndrome, etc, with active primary subfoveal, retrofoveal or juxtafoveal lesions that affect the fovea as evidenced by angiography and/or OCT in the studied eye
* Total lesion area < 12 disc areas.
* Total area of CNV within the lesion must be > 50% of total lesion.
* Best corrected visual acuity of 20/40 to 20/320 in the study eye.
* Willing and able to give informed consent.

Exclusion Criteria:

* Prior treatment in the study eye with, external-beam radiation therapy, subfoveal focal laser photocoagulation, vitrectomy, or transpupillary thermotherapy or other anti VEGF treatments,
* History of submacular surgery or other surgical intervention in the study eye, glaucoma filtration surgery, corneal transplant surgery,
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within one month preceding baseline,
* Extracapsular extraction of cataract with phacoemulsification within three months preceding baseline, or a history of post-operative complications within the last 12 months preceding baseline in the study eye (uveitis, cyclitis, etc.),
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication),
* Aphakia with absence of the posterior capsule in the study eye,
* Active intraocular inflammation (grade trace or above) in the study eye,
* Any active infection involving ocular adnexa including infectious conjunctivitis, keratitis, scleritis, endophthalmitis,
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye,
* Presence of a retinal pigment epithelial tear involving the macula in the study eye,
* Subfoveal fibrosis or atrophy in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-03 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Best Corrected Visual Acuity (BCVA)Measured by Early Treatment Diabetic Retinopathy Study (ETDRS)at every visit | From Baseline to month 12
  Compare of mean BCVA at every visit between the two groups to assess the efficacy of conbercept.

SECONDARY OUTCOMES:
Percentage of Participants Who Gained at Least 15/10/5 Letters in BCVA as Measured by ETDRS at month 12 | Baseline, month 12
Percentage of Participants Who Gained at Least 15/10/5 Letters in BCVA as Measured by ETDRS at month 6 | Baseline, month 6
Percentage of Participants Who Lost at Least 15/10/5 Letters in BCVA Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) at month 6 | Baseline, month 6
Percentage of Participants Who Lost at Least 15/10/5 Letters in BCVA Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) at month 12 | Baseline, month 12
Mean Change in Central Retinal Thickness (CRT) as Assessed by Optical Coherence Tomography (OCT) at every visit | 12 months
Mean Change in Choroidal Neovascularization (CNV) Lesion Size as Assessed by Fluorescein Angiography (FA) From Baseline to month 3/6/12 | Baseline, month 3, 6 and 12
Mean Change in European Five-dimensional Health Scale (EQ-5D) Score From Baseline to month 12 | Baseline, month 12
Mean Change in National Eye Institute 25-item Visual Function Questionnaire (NEI VFQ-25) Total Score From Baseline to month 12 | Baseline, month 12
Mean Change in Area of Leakage assessed by FFA From Baseline at month 3\6\12 | Baseline, month 3, 6 and 12
Number of participants with adverse events | 12 months
  Compare of Number of participants with adverse events between the two groups to assess the safety of conbercept

IPD SHARING:
Plan to Share IPD: Undecided